CLINICAL TRIAL: NCT06481800
Title: Progressive Muscle Relaxation Versus Manual Lymphatic Drainage on Restless Leg Syndrome and Sleep Quality in Hemodialysis Patients
Brief Title: PMR Versus MLD on RLS and Sleep Quality in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery and dermatology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005202
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Autogenic Training; Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. To assign patients to different treatment groups, a table of random numbers generated by a computer will be used. Patients will be allocated randomly into three groups using this method
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A):Progressive muscle relaxation (PMR) (Experimental): patients receive progressive muscle relaxation (PMR) for 20 minutes after each dialysis session during the first 2 hours the dialysis treatment with routine medical care for dialysis patients
  Interventions: Other: Progressive muscle relaxation (PMR)
- Group (B): Manual lymphatic drainage (MLD) (Experimental): patients receive Manual lymphatic drainage (MLD) for 20 minutes within after each dialysis session during the first 2 hours the dialysis treatment with routine medical care for dialysis patients.
  Interventions: Other: Manual lymphatic drainage (MLD)
- Group (C):control (Active Comparator): patients receive routine medical care for dialysis patients. Routine medical care for RLS and sleep quality in hemodialysis Anemia management, electrolyte balance,Avoiding caffeine and alcohol, establishing a regular sleep schedule leg care,Medicines that increase dopamine in the brain, affecting calcium channels, Opioids , Gabapentin and Pregabali , Benzodiazepines
  Interventions: Other: cnotrol group

INTERVENTIONS:
Other: Progressive muscle relaxation (PMR) — patients receive progressive muscle relaxation (PMR) for 20 minutes after each dialysis session during the first 2 hours the dialysis treatment with routine medical care for dialysis patients
  Arms: Group (A):Progressive muscle relaxation (PMR)
Other: cnotrol group — Routine medical care for RLS and sleep quality in hemodialysis Anemia management, electrolyte balance,Avoiding caffeine and alcohol, establishing a regular sleep schedule leg care,Medicines that increase dopamine in the brain, affecting calcium channels, Opioids , Gabapentin and Pregabali , Benzodiazepines,Regular monitoring of kidney function, blood tests
  Arms: Group (C):control
Other: Manual lymphatic drainage (MLD) — Manual lymphatic drainage (MLD) for 20 minutes within after each dialysis session during the first 2 hours the dialysis treatment with routine medical care for dialysis patients
  Arms: Group (B): Manual lymphatic drainage (MLD)

SUMMARY:
Progressive muscle relaxation versus manual lymphatic drainage on restless leg syndrome and sleep quality in hemodialysis patients

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) is a sensory motor disturbance with features of both neurologic and sleeps disorders. The patients complain of strong, irresistible urge to move the legs, often accompanied by uncomfortable sensations deeply in the legs. Poor sleep quality affects many hemodialysis patients and can potentially predict their morbidity, mortality, quality of life and pattern of medication use. Progressive muscle relaxation (PMR) is one way to improve physical work capacity and reduce functional limitations. Manual lymphatic drainage (MLD) is a traditional therapy in which the hands work on the tissues of the body, including tuina, acupressure, and the likes. It is beneficial to the well-being of patients both physically and mentally

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ranging from 35- 65 years old.
* Able to communicate verbally and agree to participate in the study.
* On maintenance arteriovenous fistula (AVF) hemodialysis 3 times weekly.
* None of the research participants had a lower extremity dialysis graft, and they were all taking medication to maintain their health.
* Prior to the study procedure, all patients underwent a nephrologist assessment
* All patients had good compliance with their dialysis treatment (not missing more than 2 dialysis sessions in the prior 3 months

Exclusion Criteria:

* Peripheral neuropathy or vascular diseases of the lower limbs.
* Skin diseases including acute psoriasis or eczema.
* Recent fractures or lower limbs surgeries.
* Feet injuries including severe muscle weakness, bruises, ulcers, Open wounds or recent burns

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
International restless legs syndrome rating scale (IRLS) | base line and 12 weeks.
  It consists of 10 questions considering different aspects of the impact of RLS on a patient's life. Each question can be answered with a Likert-type scale ranging from "none" (0) to "very severe" (4).
Pittsburgh Sleep Quality Index (PSQI) | base line and 12 weeks
  It is a self-report questionnaire that assesses sleep quality. The patient asked to rate his/ her sleep quality

SECONDARY OUTCOMES:
Leg cramps severity scale | base line and 12 weeks
  0 no pain (no early symptoms), 1: mild (under cramps, with early symptoms), 2: discomforting (a cramp, recovery immediate, tolerable), 3: distressing (cramps once or twice, nurse call, recover with some treatment, cramps after HD), 4: horrible and excruciating (several cramps, nurse call, not tolerable, including a cessation of HD, cramps after HD).
Patient Health Questionnaire (PHQ-9) | base line and 12 weeks
  The (PHQ-9) is efficient, reliable, and highly acceptable for diagnosing depression and anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Ahmed Abdelhady, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of progressive muscle relaxation training on anxiety levels and quality of life in dialysis patients — https://pubmed.ncbi.nlm.nih.gov/16898100/
- See also: The Effect of Progressive Relaxation Exercises on Pain, Fatigue, and Quality of Life in Dialysis Patients — https://pubmed.ncbi.nlm.nih.gov/31567304/